CLINICAL TRIAL: NCT06378710
Title: Haemodynamic and Respiratory Effects of a Low Positive End Expiratory Pressure Associated With a Fluid Challenge in Knee-chest Position- A Randomized Interventional Study
Brief Title: Haemodynamic and Respiratory Effects of a Low Positive End Expiratory Pressure Associated With a Fluid Challenge in Knee-chest Position
Acronym: OPTIPEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-0219
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Standard PEEP (at 7 cmH2o), Vt standardized between [6- 8] ml/kg theoretical ideal weight. Taking NIBP every 3 minutes.
- Optimized PEEP (Experimental): Optimized PEEP (at 2 cmH2O), filling according to VES monitoring by esophageal Doppler before reversal, Vt standardized between [6-8] ml/kg theoretical ideal weight. Taking NIBP every 3 minutes.
  Interventions: Procedure: Optimized PEEP

INTERVENTIONS:
Procedure: Optimized PEEP — Optimized PEEP
  Arms: Optimized PEEP

SUMMARY:
The genu pectoral position is a surgical position used for spine surgery. This surgical position will lead to physiological hemodynamic and respiratory changes during the procedure.

The knee-pectoral position notably induces an increase in CRF and improves pulmonary ventilation/perfusion ratios. On the other hand, it has been shown that it is accompanied by a reduction in cardiac output of approximately 15% Protective perioperative ventilation including a tidal volume between 6 and 8 ml/kg of theoretical ideal weight, PEEP and alveolar recruitment maneuvers is applied in the operating room to reduce postoperative pulmonary complications. The application of high PEEP and the performance of recruitment maneuvers induce arterial hypotension through changes in intra- and transpulmonary pressures. However, investigators hypothesize that the deleterious hemodynamic effects of PEEP seem to counterbalance its beneficial respiratory effects in this particular position.

The combination of the effects of the knee-pectoral position and protective ventilation could be potentiated and be the cause of the sometimes severe arterial hypotension observed in clinical practice. Since this position improves pulmonary ventilation perfusion ratios, the investigators hypothesized that a lower PEEP and the elimination of intraoperative recruitment maneuvers could be beneficial from a hemodynamic point of view without being deleterious in terms of perioperative pulmonary complications. An exploratory study was carried out at the CAEN University Hospital in 2021 under the name PEEP POSTURE (CLERS Agreement No. 2198 of February 17, 2021) on 90 patients aiming to collect hemodynamic and respiratory parameters in 3 surgical positions: supine decubitus, ventral decubitus , pectoral genu. No difference was found in the evolution of respiratory compliance. On the other hand, a significant drop in SBP, DBP and MAP in the pectoral position was shown compared to the supine group as well as greater vascular filling.

The investigators therefore hypothesize that a reduction in PEEP and optimization of vascular filling could help reduce the adverse effects on blood pressure linked to the surgical position.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Beneficiary of Social Security or CMU
* Surgical operation under general anesthesia requiring a knee-pectoral position
* Dated and signed informed consent

Exclusion Criteria:

* BMI > 35 kg/m²
* Hemodynamic instability before placing the knee in the pectoral position.
* ASA class IV or V
* Prolonged intervention > 2 hours
* Lack of consent
* Contraindications to the use of esophageal Doppler
* Concomitant third-party clinical trial that may induce a hemodynamic or respiratory change in the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences of a MAP | baseline
  Number of occurrences of a MAP <= 65mmHg per 3 min period occurring during the period of knee pectoral position

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No